CLINICAL TRIAL: NCT04146363
Title: A Randomized, Double-blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Lebrikizumab in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Evaluation of the Efficacy and Safety of Lebrikizumab (LY3650150) in Moderate to Severe Atopic Dermatitis (ADvocate1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17801; 2019-002932-10 (EudraCT Number); J2T-DM-KGAB (Other: Eli Lilly and Company); DRM06-AD04 (Other: Dermira, Inc.)
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2022-08-29 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Dermatitis; Dermatitis, Atopic; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases | interventions — lebrikizumab

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel group, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Induction Period (Baseline-Week 16):
  Two subcutaneous (SC) injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 until Week 14.
  Maintenance Period (Week 16-Week 52):
  Two placebo SC injections as loading dose on Week 16 and Week 18. One placebo SC injection Q2W until Week 50.
  Interventions: Other: Placebo
- Lebrikizumab 250 Q2W (Experimental): Induction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
  Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection Q2W until Week 50.
  For participants who received placebo in the Induction Period, the maintenance loading dose is:
  Two 250 mg Lebrikizumab SC injections on Week 16.
  Two 250 mg Lebrikizumab SC injections on Week 18.
  To maintain the blind, for participants who received Lebrikizumab in the Induction Period, the maintenance loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 16.
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 18.
  Interventions: Biological: Lebrikizumab; Other: Placebo
- Lebrikizumab 250 Q4W (Experimental): Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
  For participants who received placebo in the Induction Period, the maintenance loading dose is:
  Two 250 mg Lebrikizumab SC injections on Week 16.
  Two placebo injections on Week 18.
  To maintain the blind, for participants who received Lebrikizumab in the Induction Period, the maintenance loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 16.
  Two placebo injections on Week 18
  Interventions: Biological: Lebrikizumab; Other: Placebo
- Escape Arm (Lebrikizumab Q2W) (Experimental): Maintenance Period (Week 16-Week 52):
  Blinded loading doses based on prior treatment assignment will be administered, followed by one 250 mg Lebrikizumab SC injection Q2W until Week 50 in an open-label fashion.
  For participants who received placebo in the Induction Period, the loading dose is:
  Two 250 mg Lebrikizumab SC injections on Week 16.
  Two 250 mg Lebrikizumab SC injections on Week 18.
  To maintain the loading dose blind, for participants who received Lebrikizumab in the Induction Period, the loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 16. One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 18.
  For participants who do not maintain an acceptable response during the Maintenance Period and entered the Escape Arm, the loading doses will be administrated at entry and 2 weeks after entry based on the treatment assignment prior to entering escape arm.
  Interventions: Biological: Lebrikizumab; Other: Placebo

INTERVENTIONS:
Biological: Lebrikizumab — Subcutaneous injection
  Other Names: LY3650150; DRM06
  Arms: Escape Arm (Lebrikizumab Q2W); Lebrikizumab 250 Q2W; Lebrikizumab 250 Q4W
Other: Placebo — Subcutaneous Injection

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study which is 52 weeks in duration. The study is designed to confirm the safety and efficacy of lebrikizumab as monotherapy for treatment of moderate-to-severe atopic dermatitis utilizing a 16-week induction treatment period and a 36-week long-term maintenance treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults and adolescents (≥12 years and ≥40 kg)
* Chronic atopic dermatitis (according to American Academy of Dermatology Consensus Criteria) that has been present for ≥1 year before the screening visit
* Eczema Area and Severity Index (EASI) score ≥16 at the baseline visit
* Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at the baseline visit
* ≥10% body surface area (BSA) of atopic dermatitis involvement at the baseline visit
* History of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable

Exclusion Criteria:

* Prior treatment with dupilumab or tralokinumab
* Treatment with topical corticosteroids, calcineurin inhibitors or phosphodiesterase-4 inhibitors such as crisaborole within 1 week prior to the baseline visit
* Treatment with any of the following agents within 4 weeks prior to the baseline visit:

  * Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
  * Phototherapy and photochemotherapy (PUVA) for AD
* Treatment with the following prior to the baseline visit:

  * An investigational drug within 8 weeks or within 5 half-lives (if known) of baseline, whichever is longer
  * Cell-depleting biologics, including to rituximab, within 6 months of baseline
  * Other biologics within 5 half-lives (if known) or 16 weeks of baseline, whichever is longer
* Treatment with a live (attenuated) vaccine within 12 weeks of the baseline visit or planned during the study
* Uncontrolled chronic disease that might require bursts of oral corticosteroids, e.g., co-morbid severe uncontrolled asthma
* Evidence of active acute or chronic hepatitis
* History of human immunodeficiency virus (HIV) infection or positive HIV serology
* History of malignancy, including mycosis fungoides, within 5 years before the screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (94):
- United States (30):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Wallace Medical Group, Inc., Beverly Hills, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Belle Aimee Skincare Clinic, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - ACRC Studies, San Diego, California
  - Central Connecticut Dermatology, Cromwell, Connecticut
  - St. Francis Medical Institute, Clearwater, Florida
  - Community Research Foundation Inc, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - IACT Health - VHC, Columbus, Georgia
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St Joseph Dermatology and Vein Clinic, Saint Joseph, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - JDR Dermatology Research, Las Vegas, Nevada
  - ALLCUTIS Research, Portsmouth, New Hampshire
  - Icahn Sch of Med at Mt. Sinai, New York, New York
  - Sadick Research Group, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Clinical Research Institute, Medford, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Bellaire Dermatology, Bellaire, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Premier Clinical Research, Spokane, Washington
- Australia (11):
  - The St. George Hospital, Kogarah, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Skin & Cancer Foundation Australia, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Skin Health Institute Inc., Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - Burswood Dermatology, Victoria Park, Western Australia
- Canada (5):
  - CARe Clinic, Red Deer, Alberta
  - CCA Medical Research, Ajax, Ontario
  - Skin Health, Cobourg, Ontario
  - Dermatology and Dermatologic Surgery, Ottawa, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
- Kliiniliste uuringute Keskus OU, Tartu, Estonia
- France (5):
  - Hopital Saint-Louis, Paris, Cedex 10
  - CHU de Bordeaux Hopital Saint Andre, Bordeaux
  - CHU DIJON - Hopital le Bocage, Dijon
  - Cabinet Médical, Martigues
  - Hopital Larrey, Toulouse
- Latvia (5):
  - Clinic of Dermatology and STD, Riga
  - Health Center 4, Affiliate Diagnostic Center, Riga
  - Health and Aesthetics LTD, Riga
  - Latvian Dermatology Institute, Riga
  - Smite Aija - Practice in Dermatology Venereology, Talsi
- Lithuania (7):
  - JSC "CD8 Alergology Clinic", Kaunas
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Jsc Renmeda, Vilnius
  - JSC "Center for Diagnosis and Treatment of Allergic Diseases", Vilnius
  - Children's Hospital, Affiliate of Vilnius University Hospital Santaros klinikos, Vilnius
  - Inlita (Santaros CTC), Vilnius
  - Vilnius University Hospital Santaros klinikos, Vilnius
- Poland (12):
  - Diamond Clinic, Krakow, Lesser Poland Voivodeship
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp Z O.O., Tarnów, Malopolska
  - Centralny Szpital Kliniczny MSWiA, Warsaw, Masovian Voivodeship
  - Zespol Naukowo - Leczniczy "Iwolang" Sp. z o.o., Iwonicz-Zdrój, Podkarpackie Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - GynCentrum Sp z o.o., Katowice
  - Specjalistyczny Osrodek Alergologiczno-Internistyczny ALL-ME, Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Lublin
  - Centrum Alergologii Teresa Hofman, Poznan
  - Clinical Research Group Sp. z o.o., Warsaw
  - CityClinic Przychodnia Lekarsko-Psychologiczna, Wroclaw
- South Korea (11):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Pusan National University Hospital, Pusan, Korea
  - Hanyang University Medical Center, Seoul, Korea
  - Ulsan University Hospital, Ulsan, Korea
  - Ajou University Hospital, Suwon, Kyung Gi-Do, Korea
  - Soon Chun Hyang University Seoul Hospital, Seoul, Yongsan-gu
  - Incheon St. Mary's Hospital, Incheon
  - Severance Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Chungang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (7):
  - Sant Joan de Deu Serveis En Salut Mental, SANT BOI de Llobrega, Barcelona
  - Hospital De Basurto, Bilbao, Vizcaya
  - Hospital General Universitario Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Sher ER, Golant A, de Bruin-Weller M, Carrascosa JM, Mehta V, Bieber T, Dawson Z, Atwater AR, Zhong J, Rodriguez Calleja L, Boguniewicz M. Lebrikizumab is efficacious in adults and adolescents with moderate-to-severe atopic dermatitis regardless of atopic comorbidities. Ann Allergy Asthma Immunol. 2025 Dec 21:S1081-1206(25)01389-4. doi: 10.1016/j.anai.2025.12.017. Online ahead of print. PMID 41435984
- [Derived] Silverberg JI, Wollenberg A, Stein Gold L, Yosipovitch G, Lio P, Vestergaard C, Stander S, Carrascosa JM, Gallo G, Casillas M, Ding Y, Yang FE, Pierce E, Agell H, Del Rosso J. Lebrikizumab provides stable skin response with no or minimal fluctuations for up to 2 years in patients with atopic dermatitis. Clin Exp Dermatol. 2025 Nov 8:llaf490. doi: 10.1093/ced/llaf490. Online ahead of print. PMID 41206702
- [Derived] Guttman-Yassky E, Sun Z, Mena LR, Hahn N, Nickoloff BJ, Preuss C, Siu K, Natalie CR, Gallo G, Wolf E, Eyerich K, Aparici M, Benschop RJ, Okragly A. Lebrikizumab Rapidly Lowers Inflammatory Biomarkers with Clinical Correlations in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Sep;15(9):2595-2614. doi: 10.1007/s13555-025-01481-4. Epub 2025 Jul 15. PMID 40663228
- [Derived] Simpson E, Fernandez-Penas P, de Bruin-Weller M, Lio PA, Chu CY, Ezzedine K, Agell H, Casillas M, Ding Y, Yang FE, Pierce E, Bieber T. Improvement Across Dimensions of Disease with Lebrikizumab Use in Atopic Dermatitis: Two Phase 3, Randomized, Double-Blind, Placebo-Controlled Monotherapy Trials (ADvocate1 and ADvocate2). Adv Ther. 2025 Jan;42(1):132-143. doi: 10.1007/s12325-024-02974-y. Epub 2024 Sep 9. PMID 39249591
- [Derived] Silverberg JI, Wollenberg A, Stein Gold L, Del Rosso J, Yosipovitch G, Lio P, Carrascosa JM, Gallo G, Ding Y, Xu Z, Casillas M, Pierce E, Agell H, Stander S. Patients with Moderate-to-Severe Atopic Dermatitis Maintain Stable Response with No or Minimal Fluctuations with 1 Year of Lebrikizumab Treatment. Dermatol Ther (Heidelb). 2024 Aug;14(8):2249-2260. doi: 10.1007/s13555-024-01226-9. Epub 2024 Aug 10. PMID 39123054
- [Derived] Yosipovitch G, Lio P, Legat FJ, Chovatiya R, Deleuran M, Pierce E, Casillas M, Ding Y, Yang FE, Bardolet L, Stander S. Stable Response and Sustained Improvement of Itch and Sleep Symptoms in Patients with Atopic Dermatitis Treated with Lebrikizumab over 52 Weeks. Dermatol Ther (Heidelb). 2024 Aug;14(8):2171-2180. doi: 10.1007/s13555-024-01225-w. Epub 2024 Jul 13. PMID 39002092
- [Derived] Lio PA, Armstrong A, Gutermuth J, Nosbaum A, Sofen H, Gil EG, Casillas M, Chen S, Sun L, Pierce E, Elmaraghy H, Dawson Z, Torres T. Lebrikizumab Improves Quality of Life and Patient-Reported Symptoms of Anxiety and Depression in Patients with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1929-1943. doi: 10.1007/s13555-024-01199-9. Epub 2024 Jun 26. PMID 38922484
- [Derived] Simpson EL, de Bruin-Weller M, Hong HC, Staumont-Salle D, Blauvelt A, Eyerich K, Gooderham M, Shahriari M, Mallbris L, Atwater AR, Rueda MJ, Ding Y, Liu Z, Agell H, Silverberg JI. Lebrikizumab Provides Rapid Clinical Responses Across All Eczema Area and Severity Index Body Regions and Clinical Signs in Adolescents and Adults with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 May;14(5):1145-1160. doi: 10.1007/s13555-024-01158-4. Epub 2024 May 3. PMID 38700646
- [Derived] Soung J, Stander S, Gutermuth J, Pau-Charles I, Dawson Z, Yang FE, Sun L, Pierce E, Elmaraghy H, Stein-Gold L. Lebrikizumab monotherapy impacts on quality of life scores through improved itch and sleep interference in two Phase 3 trials. J Dermatolog Treat. 2024 Dec;35(1):2329240. doi: 10.1080/09546634.2024.2329240. Epub 2024 Apr 28. PMID 38679419
- [Derived] Blauvelt A, Thyssen JP, Guttman-Yassky E, Bieber T, Serra-Baldrich E, Simpson E, Rosmarin D, Elmaraghy H, Meskimen E, Natalie CR, Liu Z, Xu C, Pierce E, Morgan-Cox M, Garcia Gil E, Silverberg JI. Efficacy and safety of lebrikizumab in moderate-to-severe atopic dermatitis: 52-week results of two randomized double-blinded placebo-controlled phase III trials. Br J Dermatol. 2023 May 24;188(6):740-748. doi: 10.1093/bjd/ljad022. PMID 36994947
- [Derived] Silverberg JI, Guttman-Yassky E, Thaci D, Irvine AD, Stein Gold L, Blauvelt A, Simpson EL, Chu CY, Liu Z, Gontijo Lima R, Pillai SG, Seneschal J; ADvocate1 and ADvocate2 Investigators. Two Phase 3 Trials of Lebrikizumab for Moderate-to-Severe Atopic Dermatitis. N Engl J Med. 2023 Mar 23;388(12):1080-1091. doi: 10.1056/NEJMoa2206714. Epub 2023 Mar 15. PMID 36920778
- See also: Evaluation of the Efficacy and Safety of Lebrikizumab (LY3650150) in Moderate to Severe Atopic Dermatitis (ADvocate1) — https://trials.lillytrialguide.com/en-US/trial/6duv4kD1B48RPwp63igF1U

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who did not achieve an Investigator Global Assessment (IGA) of 0 or 1 or EASI-75 at Week 16 and those participants who did not maintain an Eczema Area and Severity Index (EASI)-50 response following re-randomization at Weeks 24, 32, 40, or 48 were assigned to an Escape Arm and received 250 mg Lebrikizumab as open-label Q2W through Week 52.
Groups:
- Induction - Placebo: Induction Period (Baseline-Week 16):
  Two subcutaneous (SC) injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 until Week 14.
- Induction - Lebrikizumab Q2W: Induction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
- Maintenance Blinded Treatment - Placebo Responder/Placebo (PBO): Maintenance Secondary Population: Maintenance Period (Week 16 to Week 52):
  One SC injection of Placebo Q2W until Week 50.
  Two placebo SC injections as loading dose on Week 16 and Week 18.
- Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q4W: Maintenance Secondary Population: Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
  For participants who received placebo in the Induction Period, the maintenance loading dose is:
  Two 250 mg Lebrikizumab SC injections on Week 16. Two placebo injections on Week 18.
- Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q2W: Maintenance Secondary Population: Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection Q2W until Week 50.
  For participants who received placebo in the Induction Period, the maintenance loading dose is:
  Two 250 mg Lebrikizumab SC injections on Week 16.
  Two 250 mg Lebrikizumab SC injections on Week 18.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo: Maintenance Primary Population: Maintenance Period (Week 16 to Week 52): One SC injection of Placebo Q2W until Week 50.
  Two placebo SC injections as loading dose on Week 16 and Week 18.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W: Maintenance Primary Population: Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
  To maintain the blind, for participants who received Lebrikizumab in the Induction Period, the maintenance loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 16.
  Two placebo injections on Week 18.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W: Maintenance Primary Population: Maintenance Period (Week 16 to Week 52):
  One 250 mg Lebrikizumab SC injection Q2W until Week 50.
  To maintain the blind, for participants who received Lebrikizumab in the Induction Period, the maintenance loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 16.
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 18.
- Escape Arm Week 16 - Maintenance Open Label - Placebo Nonresponder/ Lebrikizumab 250 Q2W: Maintenance Escape Period (Week 16 to Week 52):
  Blinded loading doses based on prior treatment assignment will be administered, followed by one 250 mg Lebrikizumab SC injection Q2W until Week 50 in an open-label fashion.
  For participants who received placebo in the Induction Period, the loading dose is:
  Two 250 mg Lebrikizumab SC injection on Week 16. Two 250 mg Lebrikizumab SC injections on Week 18.
  For participants who do not maintain an acceptable response during the Maintenance Period and entered the Escape Arm, the loading doses will be administrated at entry and 2 weeks after entry based on the treatment assignment prior to entering escape arm.
  Participants who did not achieve an EASI-50 response after 8 weeks in the Escape Arm were terminated from the study.
- Escape Arm Week 16 - Maintenance Open Label - Lebrikizumab Nonresponder/ Lebrikizumab 250 Q2W: Maintenance Escape Period (Week 16 to Week 52):
  Blinded loading doses based on prior treatment assignment will be administered, followed by one 250 mg Lebrikizumab SC injection Q2W until Week 50 in an open-label fashion.
  To maintain the loading dose blind, for participants who received Lebrikizumab in the Induction Period, the loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo on Week16. One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 18.
  For participants who do not maintain an acceptable response during the Maintenance Period and entered the Escape Arm, the loading doses will be administrated at entry and 2 weeks after entry based on the treatment assignment prior to entering escape arm.
  Participants who did not achieve an EASI-50 response after 8 weeks in the Escape Arm were terminated from the study.
- Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W: Maintenance Escape Period (Week 24 to Week 48): One 250 mg Lebrikizumab SC injection Q2W.
Period: Induction Period
Arm/Group | Induction - Placebo | Induction - Lebrikizumab Q2W | Maintenance Blinded Treatment - Placebo Responder/Placebo (PBO) | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q2W | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Lebrikizumab Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W
Started | 141 | 283 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 141 | 282 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 120 (Completed includes Responders n=24; Nonresponders n=96) | 263 (Completed includes Responders n=157; Nonresponders n=106) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 21 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Due to Epidemic/Pandemic | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Positive quantiferon test | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Blinded Treatment Period
Arm/Group | Induction - Placebo | Induction - Lebrikizumab Q2W | Maintenance Blinded Treatment - Placebo Responder/Placebo (PBO) | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q2W | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Lebrikizumab Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W
Started | 0 (Participants were assigned to this arm only during Induction Period.) | 0 (Participants were assigned to this arm only during Induction Period.) | 4 (Participants who responded to treatment, defined as and IGA of 0 or 1 or a 75% reduction in EASI from baseline to Week 16 entered the Maintenance Period and re-randomized to the following treatment groups: lebrikizumab 250 mg Q2W, lebrikizumab 250 mg Q4W, or placebo Q2W.) | 10 (Participants who responded to treatment, defined as and IGA of 0 or 1 or a 75% reduction in EASI from baseline to Week 16 entered the Maintenance Period and re-randomized to the following treatment groups: lebrikizumab 250 mg Q2W, lebrikizumab 250 mg Q4W, or placebo Q2W.) | 10 (Participants who responded to treatment, defined as and IGA of 0 or 1 or a 75% reduction in EASI from baseline to Week 16 entered the Maintenance Period and re-randomized to the following treatment groups: lebrikizumab 250 mg Q2W, lebrikizumab 250 mg Q4W, or placebo Q2W.) | 32 (Participants who responded to treatment, defined as and IGA of 0 or 1 or a 75% reduction in EASI from baseline to Week 16 entered the Maintenance Period and re-randomized to the following treatment groups: lebrikizumab 250 mg Q2W, lebrikizumab 250 mg Q4W, or placebo Q2W.) | 63 (Participants who responded to treatment, defined as and IGA of 0 or 1 or a 75% reduction in EASI from baseline to Week 16 entered the Maintenance Period and re-randomized to the following treatment groups: lebrikizumab 250 mg Q2W, lebrikizumab 250 mg Q4W, or placebo Q2W.) | 62 (Participants who responded to treatment, defined as and IGA of 0 or 1 or a 75% reduction in EASI from baseline to Week 16 entered the Maintenance Period and re-randomized to the following treatment groups: lebrikizumab 250 mg Q2W, lebrikizumab 250 mg Q4W, or placebo Q2W.) | 0 | 0 | 0
Completed | 0 | 0 | 2 | 10 | 9 | 22 | 54 | 48 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 1 | 10 | 9 | 14 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 5 | 0 | 0 | 0
Not completed — Entered Escape Arm | 0 | 0 | 1 | 0 | 0 | 7 | 4 | 6 | 0 | 0 | 0
Period: Maintenance Open Label Escape Arm
Arm/Group | Induction - Placebo | Induction - Lebrikizumab Q2W | Maintenance Blinded Treatment - Placebo Responder/Placebo (PBO) | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q2W | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Lebrikizumab Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W
Started | 0 | 0 | 0 (Maintenance period responders did not enter Maintenance Open Label Escape Arm.) | 0 (Maintenance period responders did not enter Maintenance Open Label Escape Arm.) | 0 (Maintenance period responders did not enter Maintenance Open Label Escape Arm.) | 0 (Maintenance period responders did not enter Maintenance Open Label Escape Arm.) | 0 (Maintenance period responders did not enter Maintenance Open Label Escape Arm.) | 0 (Maintenance period responders did not enter Maintenance Open Label Escape Arm.) | 96 (Only participants who did not achieve an IGA score of 0 or 1 nor an EASI-75 at Week 16 or who received any rescue therapy between Baseline to Week 16 were assigned to an Escape Arm at Week 16.) | 106 (Only participants who did not achieve an IGA score of 0 or 1 nor an EASI-75 at Week 16 or who received any rescue therapy between Baseline to Week 16 were assigned to an Escape Arm at Week 16.) | 18 (Following rerandomization at Week 16, participants not maintaining an EASI 50 response at Weeks 24, 32, 40, or 48 were assigned to an Escape Arm and received open label lebrikizumab 250 mg Q2W through Week 52.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 77 | 77 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 29 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 17 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — EASI Scoring Error | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction - Placebo | Induction - Lebrikizumab Q2W | Total
Number analyzed (Participants) | 141 | 283 | 424
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 37 | 55
  Between 18 and 65 years | 113 | 225 | 338
  >=65 years | 10 | 21 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 141 | 214
  Male | 68 | 142 | 210
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 7 | 7
  Asian | 31 | 39 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 16 | 33 | 49
  White | 93 | 196 | 289
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7 | 16 | 23
  South Korea | 13 | 21 | 34
  Latvia | 6 | 5 | 11
  United States | 62 | 128 | 190
  Poland | 25 | 56 | 81
  Australia | 13 | 26 | 39
  France | 0 | 7 | 7
  Lithuania | 7 | 11 | 18
  Spain | 4 | 9 | 13
  Estonia | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 16
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their Atopic Dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Baseline to Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. Markov Chain Monte Carlo Multiple Imputation (MCMC-MI) was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Induction Period (Baseline-Week 16):
  Two subcutaneous (SC) injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 until Week 14.
- Lebrikizumab Q2W: Induction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 283
percentage of participants | 12.7 [7.0 to 18.5] | 43.1 [37.1 to 49.0]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.7, 95% CI 2-sided [21.6 to 37.8]

2. Primary Outcome: Percentage of Participants Achieving Eczema Area And Severity Index (EASI-75) (≥75% Reduction in EASI Score) From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI-75 score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Baseline to Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 283
percentage of participants | 16.2 [9.5 to 22.8] | 58.8 [52.9 to 64.7]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 42.0, 95% CI 2-sided [33.3 to 50.6]

3. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 2
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Baseline to Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 283
percentage of participants | 0.7 [0.0 to 2.1] | 2.5 [0.7 to 4.4]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.218644, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.7, 95% CI 2-sided [-0.6 to 4.0]

4. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 4
Description: as for outcome 3
Time Frame: Baseline to Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 283
percentage of participants | 0.8 [-0.7 to 2.3] | 10.6 [6.9 to 14.2]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000498, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.6, 95% CI 2-sided [5.7 to 13.6]

5. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 16 in Adults
Description: as for outcome 3
Time Frame: Baseline to Week 16
Population: All randomized adult participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 123 | 246
percentage of participants | 11.3 [5.4 to 17.2] | 42.2 [35.8 to 48.6]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 30.8, 95% CI 2-sided [22.1 to 39.4]

6. Secondary Outcome: Percentage of Participants Achieving EASI-90 (≥90% Reduction in EASI Score) From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-90 responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the EASI score.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 283
percentage of participants | 9.0 [3.9 to 14.0] | 38.3 [32.5 to 44.1]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.8, 95% CI 2-sided [21.3 to 36.3]

7. Secondary Outcome: Percent Change in Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable." Least Squares (LS) Mean was calculated using analysis of covariance (ANCOVA) model with treatment and randomization strata (region, disease severity, age) as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with a Baseline Pruritus NRS score >0, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 136 | 276
percent change | -15.06 (3.833) | -45.48 (3.143)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -30.42, 95% CI 2-sided [-38.1 to -22.7], Standard Error of Mean 3.915

8. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥4-points at Baseline Who Achieve a ≥4-point Reduction in Pruritus NRS Score From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Time Frame: Baseline to Week 16
Population: All randomized participants, with a Baseline Pruritus NRS score ≥4, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 130 | 263
percentage of participants | 13.0 [7.0 to 18.9] | 45.9 [39.8 to 52.1]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 32.9, 95% CI 2-sided [24.6 to 41.3]

9. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥5-points at Baseline Who Achieve a ≥4-point Reduction in Pruritus NRS Score From Baseline to Week 16
Description: as for outcome 8
Time Frame: Baseline to Week 16
Population: All randomized participants, with Baseline Pruritus NRS score ≥ 5, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 123 | 244
percentage of participants | 13.7 [7.5 to 20.0] | 49.0 [42.7 to 55.4]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 35.1, 95% CI 2-sided [26.3 to 43.9]

10. Secondary Outcome: Percent Change in EASI Score From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  LS Mean was calculated using ANCOVA model with treatment, stratification factors of geographic region, age group, baseline IGA score (IGA 3 versus 4) as fixed factors baseline value as covariate.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 283
percent change | -26.01 (4.031) | -64.31 (3.156)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -38.31, 95% CI 2-sided [-46.4 to -30.2], Standard Error of Mean 4.151

11. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) at Week 16
Description: The BSA affected by AD will be assessed for 4 separate body regions: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. BSA was calculated using the participant's palm using the 1% rule, 1 palm was equivalent to 1% with estimates of the number of palms it takes to cover the affected AD area. Maximum number of palms were 10 palms for head and neck (10%), 20 palms for upper extremities (20%), 30 palms for trunk, including axilla and groin (30%), 40 palms for lower extremities, including buttocks (40%). Percent of BSA for a body region was calculated as = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA of all 4 body regions ranges from 0% to 100 % with higher values representing greater severity of AD.
Time Frame: Baseline, Week 16
Population: All randomized participants, with observed BSA data, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. The mixed model repeated measures (MMRM) included treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit, geographic region, age group, baseline IGA score. MMRM was used to handle all missing data.
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 77 | 235
percentage of body surface area | -11.7 (1.86) | -30.2 (1.31)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Mixed Models Analysis; LS Mean Difference (Final Values) = -18.5, 95% CI 2-sided [-22.4 to -14.5], Standard Error of Mean 2.00

12. Secondary Outcome: Percentage of Participants Achieving EASI-90 From Baseline to Week 4
Description: as for outcome 6
Time Frame: Baseline to Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 283
percentage of participants | 1.6 [-0.6 to 3.8] | 12.4 [8.5 to 16.3]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000412, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.7, 95% CI 2-sided [6.2 to 15.2]

13. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
  LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing baseline DLQI score, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 121 | 239
score on a scale | -2.9 (1.10) | -8.7 (1.05)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-7.1 to -4.5], Standard Error of Mean 0.68

14. Secondary Outcome: Percentage of Participants Achieving ≥4 Point Improvement in DLQI From Baseline to Week 16
Description: The DLQI is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
Time Frame: Baseline to Week 16
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 121 | 239
percentage of participants | 32.4 [23.8 to 41.1] | 71.5 [65.7 to 77.4]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 38.8, 95% CI 2-sided [28.3 to 49.3]

15. Secondary Outcome: Percentage of Participants With a DLQI Total Score of ≥4-point at Baseline Achieving ≥4-point Improvement in DLQI From Baseline to Week 16
Description: as for outcome 14
Time Frame: Baseline to Week 16
Population: All randomized participants, with a DLQI Total Score of ≥4-point at baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 116 | 226
percentage of participants | 33.8 [24.9 to 42.8] | 75.6 [69.9 to 81.4]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 41.8, 95% CI 2-sided [31.2 to 52.3]

16. Secondary Outcome: Percent Change in Sleep-loss Score From Baseline to Week 16
Description: Sleep Loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all)]. Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant using an electronic diary. LS Mean was calculated using ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants, with baseline sleep-loss score >0, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 132 | 269
percent change | -15.99 (5.139) | -48.33 (4.175)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -32.35, 95% CI 2-sided [-42.6 to -22.1], Standard Error of Mean 5.230

17. Secondary Outcome: Change From Baseline in Sleep-loss Score at Week 16
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: All randomized participants, non-missing baseline Sleep-loss score, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 136 | 276
score on a scale | -0.38 (0.096) | -1.13 (0.078)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-0.9 to -0.6], Standard Error of Mean 0.098

18. Secondary Outcome: Percentage of Participants With a Sleep-loss Score ≥2 Points at Baseline Who Achieve a ≥2 Points Reduction From Baseline at Week 16
Description: Sleep Loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all)]. Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant using an electronic diary.
Time Frame: Baseline to Week 16
Population: All randomized participants, with baseline sleep-loss score ≥2 Points, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 91 | 195
percentage of participants | 4.7 [0.3 to 9.2] | 39.0 [32.1 to 46.0]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 34.6, 95% CI 2-sided [26.2 to 43.0]

19. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥4 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 1
Description: as for outcome 8
Time Frame: Baseline to Week 1
Population: All randomized participants, with a Pruritus NRS Score of ≥4 Points at Baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 130 | 263
percentage of participants | 0.8 [0.0 to 2.3] | 2.3 [0.5 to 4.1]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.275529, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.5, 95% CI 2-sided [-0.8 to 3.9]

20. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥4 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 2
Description: as for outcome 8
Time Frame: Baseline to Week 2
Population: All randomized participant, with a Pruritus NRS Score of ≥4 Points at Baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 130 | 263
percentage of participants | 0.9 [-0.8 to 2.5] | 6.1 [3.2 to 9.0]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.016656, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.3, 95% CI 2-sided [1.9 to 8.6]

21. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥4 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 4
Description: as for outcome 8
Time Frame: Baseline to Week 4
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 130 | 263
percentage of participants | 2.3 [0.0 to 4.9] | 21.5 [16.5 to 26.5]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000003, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.3, 95% CI 2-sided [13.7 to 25.0]

22. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥5 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 1
Description: as for outcome 8
Time Frame: Baseline to Week 1
Population: All randomized participants, with a Pruritus NRS Score of ≥5 Points at Baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 123 | 244
percentage of participants | 0.8 [0.0 to 2.4] | 2.5 [0.5 to 4.4]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.244105, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.8, 95% CI 2-sided [-0.8 to 4.3]

23. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥5 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 2
Description: as for outcome 8
Time Frame: Baseline to Week 2
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 123 | 244
percentage of participants | 0.9 [-0.9 to 2.7] | 6.6 [3.5 to 9.7]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.014450, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.8, 95% CI 2-sided [2.2 to 9.4]

24. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥5 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 4
Description: as for outcome 8
Time Frame: Baseline to Week 4
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 123 | 244
percentage of participants | 2.4 [0.0 to 5.2] | 23.1 [17.8 to 28.5]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.9, 95% CI 2-sided [14.9 to 26.9]

25. Secondary Outcome: Percent Change in SCORing Atopic Dermatitis (SCORAD) From Baseline to Week 16
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  LS Mean was calculated using the ANCOVA model with treatment group and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with baseline SCORAD >0, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. Missing Values were imputed using last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 138 | 276
percent change | -16.64 (3.162) | -46.93 (2.551)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -30.29, 95% CI 2-sided [-36.59 to -24.00], Standard Error of Mean 3.203

26. Secondary Outcome: Pharmacokinetics (PK): Average Serum Concentration of Lebrikizumab at Week 52
Description: PK: Average serum concentration of lebrikizumab at the Week 52 trough timepoint. Serum concentration is a combined measure obtained from Baseline, Week 4, Week 16, Week 32, Week 52 and average measure was reported at week 52.
Time Frame: Predose: Baseline, Week 4, Week 16, Week 32, Week 52
Population: All participants who were randomly assigned to lebrikizumab 250 mg Q2W at Baseline visit and randomly reassigned to lebrikizumab 250 mg Q2W, lebrikizumab 250 mg Q4W, or placebo at Week 16 and had evaluable PK data at Week 52. The 250 mg Q2W PK population also includes any placebo participants entering the Escape Arm at W16 and participants in the Maintenance Period entering the Escape Arm from 250 mg Q2W dosing.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)
Groups:
- Maintenance 250 mg Lebrikizumab Q4W: 250 mg Lebrikizumab administered SC injection Q4W.
- Maintenance 250 mg Lebrikizumab Q2W and 250 mg Lebrikizumab Escape Q2W: 250 mg Lebrikizumab administered SC injection Q2W.
Arm/Group | Maintenance 250 mg Lebrikizumab Q4W | Maintenance 250 mg Lebrikizumab Q2W and 250 mg Lebrikizumab Escape Q2W
Number analyzed (Participants) | 51 | 195
micrograms per milliliter (ug/mL) | 40.7 (23.7) | 75.7 (39.0)

27. Secondary Outcome: Percentage of Participants From Those Re-randomized Having Achieved EASI-75 at Week 16 Who Continued to Exhibit EASI-75 at Week 52 (EASI-75 Calculated Relative to Baseline EASI Score)
Description: as for outcome 2
Time Frame: Baseline to Week 52
Population: All participants who were randomized to Lebrikizumab 250 mg Q2W at Baseline Visit and re-randomized to Lebrikizumab 250 mg Q2W, Lebrikizumab 250 mg Q4W or placebo at Week 16 and received at least 1 dose of study treatment during the maintenance period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo: Participants received placebo administered SC injection Q2W.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W: Participants received 250 mg Lebrikizumab administered SC injection Q4W.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W: Participants received 250 mg Lebrikizumab administered SC injection Q2W.
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 30 | 62 | 61
percentage of participants | 61.3 [42.3 to 80.4] | 79.2 [68.0 to 90.4] | 79.2 [67.6 to 90.8]
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.072375, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.9, 95% CI 2-sided [-2.3 to 38.1]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.106653, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.5, 95% CI 2-sided [-4.5 to 39.5]

28. Secondary Outcome: Percentage of Participants From Those Re-randomized Having Achieved IGA 0 or 1 and a ≥2-point Improvement From Baseline at Week 16 Who Continue to Exhibit and IGA 0 or 1 and a ≥2-point Improvement From Baseline at Week 52
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 22 | 45 | 45
percentage of participants | 46.5 [24.4 to 68.7] | 74.2 [60.5 to 88.0] | 75.8 [62.9 to 88.7]
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.029857, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.0, 95% CI 2-sided [2.8 to 53.2]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.019744, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.0, 95% CI 2-sided [4.6 to 53.3]

29. Secondary Outcome: Percentage of Participants From Those With a Pruritus NRS of ≥4-points at Baseline Re-randomized Having Achieved ≥4-point Reduction From Baseline at Week 16 Who Continue to Exhibit ≥4-point Reduction From Baseline at Week 52
Description: as for outcome 8
Time Frame: Baseline to Week 52
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 17 | 29 | 38
percentage of participants | 65.4 [41.5 to 89.3] | 80.4 [63.5 to 97.3] | 81.2 [68.0 to 94.3]
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.268265, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.8, 95% CI 2-sided [-12.2 to 43.8]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.192776, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.6, 95% CI 2-sided [-9.4 to 42.7]

30. Secondary Outcome: Percentage of Participants From Those With a Pruritus NRS of ≥5-points at Baseline Re-randomized Having Achieved ≥4-point Reduction From Baseline at Week 16 Who Continue to Exhibit ≥4-point Reduction From Baseline at Week 52
Description: as for outcome 8
Time Frame: Baseline to Week 52
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 17 | 28 | 38
percentage of participants | 65.4 [41.5 to 89.3] | 83.3 [66.7 to 99.9] | 81.2 [68.0 to 94.3]
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.185361, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.6, 95% CI 2-sided [-9.3 to 46.6]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.192776, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.6, 95% CI 2-sided [-9.4 to 42.7]

31. Secondary Outcome: Percent Change in SCORAD (Having Achieved EASI-75 at Week 16) From Baseline at Week 52
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. LS mean was calculated using ANCOVA model with treatment group, baseline value, and stratification factors geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 52
Population: All participants who were randomized to Lebrikizumab 250 mg Q2W at Baseline Visit and re-randomized to Lebrikizumab 250 mg Q2W, Lebrikizumab 250 mg Q4W or placebo at Week 16 and received at least 1 dose of study treatment during the maintenance period. Missing Values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 29 | 59 | 60
percent change | -69.65 (3.972) | -71.39 (2.870) | -75.28 (2.818)
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.714208, ANCOVA; LS Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-11.15 to 7.66], Standard Error of Mean 4.756
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.237855, ANCOVA; LS Mean Difference (Final Values) = -5.63, 95% CI 2-sided [-15.01 to 3.76], Standard Error of Mean 4.4748

32. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) at Week 16 - Health State Index
Description: The EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1, with higher score indicating better health state.
  LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing EQ-5D-5L data at baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. Missing Values were imputed using last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Lebrikizumab Q2W: Induction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
  .
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 282
score on a scale
  Health State Index UK | 0.0 (0.02) | 0.2 (0.01)
  Health State Index US | 0.0 (0.01) | 0.1 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; UK; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = 0.1, 95% CI 2-sided [0.1 to 0.2], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Placebo vs Lebrikizumab Q2W; US; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = 0.1, 95% CI 2-sided [0.1 to 0.1], Standard Error of Mean 0.01

33. Secondary Outcome: Change From Baseline in EQ-5D-5L at Week 16 - Visual Analog Scale (VAS)
Description: The EQ-5D-5L is a 2-part measurement. The second part is assessed using a VAS that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine. LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing EQ-5D-5L data at baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 282
score on a scale | 2.1 (1.64) | 10.4 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = 8.3, 95% CI 2-sided [5.0 to 11.5], Standard Error of Mean 1.66

34. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) at Week 16
Description: POEM is a 7-item, validated, questionnaire used by the participant to assess disease symptoms over the last week. The participant is asked to respond to 7 questions on skin dryness, itching, flaking, cracking, sleep loss, bleeding and weeping. All 7 answers carry equal weight with a total possible score from 0 to 28 (answers scored as: No days=0; 1# 2 days = 1; 3-4 days = 2; 5#6 days = 3; everyday = 4). A high score is indicative of a poor quality of life. POEM responses will be captured using an electronic diary and transferred into the clinical database. LS Mean was calculated using MMRM model using treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit as covariates, geographic region, age group, baseline IGA (3 versus 4) score as fixed.
Time Frame: Baseline, Week 16
Population: All randomized participants, with observed POEM data, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MMRM was used to handle all missing data
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 71 | 205
score on a scale | -3.9 (0.72) | -11.3 (0.47)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Mixed Models Analysis; LS Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-8.9 to -5.7], Standard Error of Mean 0.80

35. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety at Week 16 - Adolescents
Description: PROMIS® is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Participants ≤17 years will complete pediatric versions for the duration of the study. PROMIS anxiety has 8 questions on Emotion Distress-Anxiety (or Pediatric Anxiety Symptom). Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-Scores (mean = 50 and a standard deviation = 10) with higher scores representing greater anxiety. LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized, adolescent participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 18 | 37
T-score | -2.80 (2.435) | -3.87 (1.830)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.716224, ANCOVA; LS Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-6.93 to 4.80], Standard Error of Mean 2.917

36. Secondary Outcome: Change From Baseline in PROMIS Depression at Week 16 - Adolescents
Description: PROMIS® is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Participants ≤17 years will complete pediatric versions for the duration of the study. PROMIS depression has 8 questions on Emotion Distress-Depression (or Pediatric Depressive Symptom). Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-Scores (mean = 50 and a standard deviation = 10) with higher scores representing greater depression. LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: as for outcome 35
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 18 | 37
T-score | -0.11 (2.165) | -4.62 (1.623)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.089275, ANCOVA; LS Mean Difference (Final Values) = -4.51, 95% CI 2-sided [-9.73 to 0.72], Standard Error of Mean 2.599

37. Secondary Outcome: Change From Baseline in PROMIS Anxiety at Week 16 - Adults
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The PROMIS measures will be completed by the participant in the study clinic. PROMIS anxiety has 8 questions on Emotion Distress-Anxiety (or Pediatric Anxiety Symptom). Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-Scores (mean = 50 and a standard deviation = 10) with higher scores representing greater anxiety. LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized, adults participants, with Week 16 PROMIS anxiety data, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. Missing Values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 122 | 244
T-score | -0.60 (0.660) | -3.91 (0.475)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000040, ANCOVA; LS Mean Difference (Final Values) = -3.31, 95% CI 2-sided [-4.88 to -1.75], Standard Error of Mean 0.796

38. Secondary Outcome: Change From Baseline in PROMIS Depression at Week 16 - Adults
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The PROMIS measures will be completed by the participant in the study clinic. PROMIS depression has 8 questions on Emotion Distress-Depression (or Pediatric Depressive Symptom). Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-Scores (mean = 50 and a standard deviation = 10) with higher scores representing greater depression. LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized, adult participants, with Week 16 PROMIS Depression data, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 122 | 244
T-score | -0.37 (0.579) | -3.07 (0.416)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000127, ANCOVA; LS Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-4.07 to -1.33], Standard Error of Mean 0.697

39. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) Score at Week 16 in Participants Who Have Self-Reported Comorbid Asthma
Description: The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/ limitation) scale. The ACQ-5 score is the average of the individual item scores and ranges from 0 (totally controlled) to 6 (severely uncontrolled). Higher scores indicate lower asthma control.
  LS Mean was calculated using ANCOVA with treatment, geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing baseline ACQ-5 score, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 51 | 95
score on a scale | -0.05 (0.117) | -0.14 (0.095)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.455291, ANCOVA; LS Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.33 to 0.15], Standard Error of Mean 0.121

40. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) at Week 16 - Adolescents
Description: The CDLQI questionnaire is designed for use in children (4 to 16 years of age). It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. The scoring of each question is: Very much =3; Quite a lot = 2; Only a little = 1; Not at all = 0. CDLQI total score is calculated by summing all 10 items responses and has a range of 0 to 30 (higher scores are indicative of greater impairment).
  LS Mean was calculated using MMRM model which includes treatment, baseline value, visit, the interaction of the baseline value-by-visit as covariates, the interaction of treatment by-visit, geographic region, age group, and baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized, adolescent participants, with non-missing baseline CDLQI score, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MMRM was used to handle all missing data
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 9 | 26
score on a scale | -1.0 (1.29) | -8.0 (0.80)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000069, Mixed Models Analysis; LS Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-10.1 to -3.9], Standard Error of Mean 1.52

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Induction - Lebrikizumab 250mg Q2W: IInduction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
- Maintenance Blinded - Lebrikizumab Responder/ Placebo: Maintenance Period (Week 16 to Week 52): One 250 mg SC injection of Placebo Q2W.
- Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q4W: Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection and one placebo SC injection as maintenance loading dose on Week 16 and two placebo SC injections on Week 18.
  One 250 mg Lebrikizumab SC injection Every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
- Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q2W; Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W: Maintenance Period (Week 16 to Week 52): One 250 mg Lebrikizumab SC injection Q2W.
- Maintenance Blinded - Placebo Responder/ Placebo: Maintenance Period (Week 16 to Week 52): One SC injection of Placebo Q2W.
- Maintenance Blinded - Placebo Responder/Lebrikizumab Q4W: Maintenance Period (Week 16 to Week 52):
  One 250 mg Lebrikizumab SC injection and one placebo SC injection as maintenance loading dose on Week 16 and two placebo SC injections on Week 18.
  One 250 mg Lebrikizumab SC injection Every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
- Escape Arm Week 16 - Maintenance Open Label (OL) -Placebo Non-Responder/Lebrikizumab Q2W: Maintenance Escape Period (Week 16 to Week 52): One 250 mg Lebrikizumab SC injection Q2W.
- Escape Arm Week 16 - Maintenance OL- Lebrikizumab Non-Responder/Lebrikizumab Q2W: Maintenance Escape Period (Week 16to Week 52): One 250 mg Lebrikizumab SC injection Q2W.
- Escape Arm Week 24 to 48 - Maintenance Lebrikizumab: Maintenance Escape Period (Week 24 to Week 48): One 250 mg Lebrikizumab SC injection Q2W.
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250mg Q2W | Maintenance Blinded - Lebrikizumab Responder/ Placebo | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q4W | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q2W | Maintenance Blinded - Placebo Responder/ Placebo | Maintenance Blinded - Placebo Responder/Lebrikizumab Q4W | Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W | Escape Arm Week 16 - Maintenance Open Label (OL) -Placebo Non-Responder/Lebrikizumab Q2W | Escape Arm Week 16 - Maintenance OL- Lebrikizumab Non-Responder/Lebrikizumab Q2W | Escape Arm Week 24 to 48 - Maintenance Lebrikizumab
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/282 | 0/32 | 0/63 | 0/62 | 0/4 | 0/10 | 0/10 | 0/96 | 0/106 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/141 | 6/282 | 0/32 | 2/63 | 0/62 | 1/4 | 0/10 | 0/10 | 1/96 | 4/106 | 0/18
Other Adverse Events (participants affected / at risk) | 73/141 | 127/282 | 15/32 | 32/63 | 25/62 | 2/4 | 4/10 | 3/10 | 51/96 | 47/106 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction - Placebo (N=141) | Induction - Lebrikizumab 250mg Q2W (N=282) | Maintenance Blinded - Lebrikizumab Responder/ Placebo (N=32) | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q4W (N=63) | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q2W (N=62) | Maintenance Blinded - Placebo Responder/ Placebo (N=4) | Maintenance Blinded - Placebo Responder/Lebrikizumab Q4W (N=10) | Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W (N=10) | Escape Arm Week 16 - Maintenance Open Label (OL) -Placebo Non-Responder/Lebrikizumab Q2W (N=96) | Escape Arm Week 16 - Maintenance OL- Lebrikizumab Non-Responder/Lebrikizumab Q2W (N=106) | Escape Arm Week 24 to 48 - Maintenance Lebrikizumab (N=18)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/73 (0) | 0/141 (0) | 0/21 (0) | 0/38 (0) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 0/45 (0) | 1/43 (1) | 0/5 (0)
Micromastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction - Placebo (N=141) | Induction - Lebrikizumab 250mg Q2W (N=282) | Maintenance Blinded - Lebrikizumab Responder/ Placebo (N=32) | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q4W (N=63) | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q2W (N=62) | Maintenance Blinded - Placebo Responder/ Placebo (N=4) | Maintenance Blinded - Placebo Responder/Lebrikizumab Q4W (N=10) | Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W (N=10) | Escape Arm Week 16 - Maintenance Open Label (OL) -Placebo Non-Responder/Lebrikizumab Q2W (N=96) | Escape Arm Week 16 - Maintenance OL- Lebrikizumab Non-Responder/Lebrikizumab Q2W (N=106) | Escape Arm Week 24 to 48 - Maintenance Lebrikizumab (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Erythropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 7 (7) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 5 (5) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucomatocyclitic crises (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoconus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pupils unequal (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vernal keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0/73 (0) | 1/141 (1) | 0/21 (0) | 0/38 (0) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 1/45 (1) | 0/43 (0) | 0/5 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 4 (4) | 21 (23) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 5 (6) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 8 (9) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecthyma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 11 (11) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (5) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 5 (10) | 9 (9) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 1/73 (1) | 0/141 (0) | 0/21 (0) | 0/38 (0) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 0/45 (0) | 0/43 (0) | 0/5 (0)
Viral pericarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/73 (0) | 2/141 (2) | 0/21 (0) | 1/38 (1) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 0/45 (0) | 0/43 (0) | 0/5 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte morphology abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nitrite urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 0/73 (0) | 0/141 (0) | 0/21 (0) | 0/38 (0) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 1/45 (1) | 0/43 (0) | 0/5 (0)
Strongyloides test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cutaneous t-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Histiocytic necrotising lymphadenitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/68 (0) | 0/141 (0) | 0/11 (0) | 0/25 (0) | 0/34 (0) | 0/2 (0) | 0/4 (0) | 0/6 (0) | 0/51 (0) | 1/63 (1) | 0/13 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 9 (10) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/68 (0) | 0/141 (0) | 0/11 (0) | 1/25 (1) | 0/34 (0) | 0/2 (0) | 0/4 (0) | 0/6 (0) | 1/51 (1) | 0/63 (0) | 0/13 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/73 (0) | 0/141 (0) | 0/21 (0) | 0/38 (0) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 1/45 (1) | 0/43 (0) | 0/5 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/73 (0) | 3/141 (5) | 0/21 (0) | 0/38 (0) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 0/45 (0) | 1/43 (4) | 0/5 (0)
Galactorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0/73 (0) | 1/141 (1) | 0/21 (0) | 0/38 (0) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 0/45 (0) | 0/43 (0) | 0/5 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/73 (0) | 0/141 (0) | 0/21 (0) | 0/38 (0) | 0/28 (0) | 0/2 (0) | 0/6 (0) | 0/4 (0) | 0/45 (0) | 1/43 (1) | 0/5 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 30 (33) | 16 (17) | 4 (4) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 4 (5) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT04146363/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT04146363/SAP_001.pdf